CLINICAL TRIAL: NCT02196896
Title: Enhancing Inpatient Psychotherapeutic Treatment With Online Self Help in a Randomised Controlled Trial: Acceptance and Efficacy
Brief Title: Enhancing Inpatient Psychotherapeutic Treatment With Online Self-help : Acceptance and Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Rhön-Klinikum AG (Unknown)
Responsible Party: Principal Investigator, M.E. Beutel, Prof. Dr., Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RK-97880
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- deprexis® (Experimental): Patients in this arm use deprexis® as an additional treatment during their inpatient stay and as an aftercare intervention.
  Interventions: Other: deprexis®
- Information (Placebo Comparator): Patients in this arm receive online information about depression as a placebo comparator in addition to their treatment during their inpatient stay and as an aftercare intervention.
  Interventions: Other: Information

INTERVENTIONS:
Other: deprexis® — Online self-help program in addition to inpatient psychosomatic treatment for 90 days.
  Arms: deprexis®
Other: Information — The patients receive online information about depression once a week for 90 days.
  Arms: Information

SUMMARY:
The purpose of this study is to determine the acceptance and efficacy of the online self-help program deprexis® for depressed patients in reducing the clinical symptoms of their depression. The patients of the experimental group use deprexis® for 90 days, the patients of the placebo group receive weekly online information about depression for 90 days as well. Both groups receive their treatment in addition to their regular inpatient psychosomatic treatment and as an aftercare intervention.The investigators hypothesize that the online self-help group achieves a greater reduction of depression compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient treatment
* Private internet access
* Informed consent
* Age between 18 and 65 years
* Knowledge of the German language
* Score in the BDI-II > 13 and clinical diagnosis of a depression (ICD-10: F32.x, F33.x, F34.1, F43.2) verified by the inpatient therapist

Exclusion Criteria:

* Psychosis
* Current alcohol or drug dependency
* Borderline, antisocial, schizoid or schizotypal personality disorder
* Anorexia nervosa
* Life time diagnosis of a schizophrenia, schizoaffective , bipolar oder organic psychic disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2014-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Reduction of depression measured with the "Beck's Depression Inventory" (BDI-II) | Three months after randomization

SECONDARY OUTCOMES:
Reduction of depression measured with the depression scale of the "Patient Health Questionnaire" (PHQ-9) | Randomization, end of inpatient treatment (average 6 weeks), six months after randomization
Reduction of depression measured with the "Beck's Depression Inventory" (BDI-II) | Randomization, end of inpatient treatment (average 6 weeks), six months after randomization
Reduction of anxiety measured with the "Generalized Anxiety Disorder Scale" (GAD-7) | Randomization, end of inpatient treatment (average 6 weeks), six months after randomization
Reduction of dysfunctional depression related cognitions measured with the "Dysfunctional Attitude Scale" (DAS) | Randomization, end of inpatient treatment (average 6 weeks), six months after randomization
Improved self-esteem measured with the "Rosenberg Self-Esteem Scale" (RSE) | Randomization, end of inpatient treatment (average 6 weeks), six months after randomization
Improved quality of life measured with the "European Health Interview Survey Quality of Life-8" (EUROHIS-QOL 8) | Randomization, end of inpatient treatment (average 6 weeks), six months after randomization
Improved working ability measured with the short form of the "Work Ability Index" (WAI) | Randomization, end of inpatient treatment (average 6 weeks), six months after randomization
Acceptance and utilization of deprexis® measured with a self devised questionnaire | End of inpatient treatment (average 6 weeks), three months after randomization
Acceptance and utilization of the information used in the placebo condition measured with a self devised questionnaire | End of inpatient treatment (average 6 weeks), three months after randomization
Degree of childhood traumas measured with the "Childhood Trauma Questionnaire" (CTQ) | Randomization
  Assumption that childhood traumas, assessed at the beginning of treatment, have a moderating effect on the reduction in the primary outcome measure.
Degree of structural deficits measured with the short form of the OPD-Structure Questionnaire (OPD-SFK) | Randomization
  Assumption that structural deficits, as assessed with the OPD-SFK questionnaire at the beginning of treatment have a moderating effect on the reduction in the primary outcome measure.
Therapeutic alliance between participant and inpatient psychotherapist measured with the "Helping Alliance Questionnaire" (HAQ). | Randomization, end of inpatient treatment (average 6 weeks)
Course of mood, depressiveness and utilization of units | During inpatient treatment (average 6 weeks)
Utilization of other treatments after the end of inpatient treatment | Six months after randomization
Satisfaction with inpatient treatment | End of inpatient treatment (average 6 weeks)
Willingness to pay | Three months after randomization
Remission from depression | End of inpatient treatment (average 6 weeks), three months after randomization, six months after randomization
  BDI score below the cutoff of 13 and a reliable change regarding Reliable Change Index (RCI)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred E Beutel, Prof. Dr., Principal Investigator — University Medical Center, Department of Psychosomatic Medicine and Psychotherapy, Johannes Gutenberg University Mainz
Locations (2):
- Germany (2):
  - Psychosomatic Clinic Bad Neustadt, Bad Neustadt an der Saale, Bavaria
  - University Medical Center, Department of Psychosomatic Medicine and Psychotherapy, Johannes Gutenberg University, Mainz, Rhineland-Palatinate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zwerenz R, Baumgarten C, Becker J, Tibubos A, Siepmann M, Knickenberg RJ, Beutel ME. Improving the Course of Depressive Symptoms After Inpatient Psychotherapy Using Adjunct Web-Based Self-Help: Follow-Up Results of a Randomized Controlled Trial. J Med Internet Res. 2019 Oct 24;21(10):e13655. doi: 10.2196/13655. PMID 31651403
- [Derived] Zwerenz R, Becker J, Knickenberg RJ, Hagen K, Dreier M, Wolfling K, Beutel ME. Enhancing inpatient psychotherapeutic treatment with online self-help: study protocol for a randomized controlled trial. Trials. 2015 Mar 17;16:98. doi: 10.1186/s13063-015-0620-6. PMID 25872505